CLINICAL TRIAL: NCT00124774
Title: Nucleoplasty for Contained Herniated Lumbar Discs: A Randomised, Double Blind, Prospective Comparison With Sham Treatment
Brief Title: Nucleoplasty for Contained Herniated Lumbar Discs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: Maastricht University (Other); ArthroCare Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-269
Record Dates: First submitted 2005-07-27; First posted 2005-07-28 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Herniated Disc
Keywords: hernia; nucleoplasty; radicular pain; Contained lumbar herniated disc
MeSH Terms: conditions — Intervertebral Disc Displacement; Hernia

INTERVENTIONS:
Procedure: Nucleoplasty

SUMMARY:
This is a prospective randomised double blind comparison trial. Fifty patients will be included, 25 in the nucleoplasty treatment group, 25 in the control group. The nucleoplasty group will undergo the nucleoplasty treatment. Control group will undergo a sham treatment. Both groups will undergo a standardised post-operative care program. The study hypothesis is that nucleoplasty will lead to earlier pain reduction as compared with the sham treatment.

DETAILED DESCRIPTION:
This study will include patients with a contained lumbar hernia of at least 6 weeks existence in whom leg pain is the predominant complaint. Standard treatment for these patients is conservative, as an operation is not without risks and is not always effective. Furthermore, complaints will usually resolve in due time. However, the pain limits the patients in their daily activities, often for a prolonged period.

In this study, nucleoplasty will be compared with a sham treatment and not with conservative treatment, as the discography is thought to have some therapeutic effect.

The primary outcome will be the proportion of patients with at least a 2.5 points decrease on a ten-point Jensen VAS score 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Mono radicular leg pain for at least 6 weeks as a result from a lumbar contained herniated disc. Leg pain must be of greater impact than concomitant back-pain
* Failing conservative treatment; analgesics and/or physical therapy. Failing means persisting pain leading to problems with daily activities.
* Magnetic resonance imaging (MRI): must be performed < 6 weeks before start treatment. On MRI signs of contained herniated disc, maximum 33% obliteration of the spinal channel. No signs of other significant spine pathology (see exclusion criteria).
* Neurological investigation by neurologist. Symptoms should be clinically related to the disc herniation level.
* Age >18 and < 60 years
* Mean leg pain on visual analogue scale (VAS) >50 mm (0 -100)

Exclusion Criteria:

* Herniated disc with more than 33% obliteration of the spinal channel.
* Annulus rupture with sequestrated herniated disc.
* Pain on VAS below 50 mm
* Pain existing longer than one year
* Less than 50% preserved disc height
* Conflict with social security/insurance.
* Major motor impairment as a result of the herniation, paresis grade 3 or more using a Medical Research Council (MRC) score
* Other degenerative causes of nerve root compression; ligament flavum or facet joint hypertrophy, degenerative spinal channel stenosis, loss of lumbar kyphosis, discopathy with signs of Schmorls' nodules and loss of nucleus pulposus signal. Other causes of radicular syndrome such as cancer, radiculitis or neural degeneration.
* Spinal instability (spondylolisthesis, spinal fracture or tumor)
* History of back surgery, chemonucleolysis or other intra discal procedures
* Coagulopathies or oral anti-coagulation therapy
* Infection
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-11; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Decrease in Jensen visual analogue scale (VAS)-score for pain

SECONDARY OUTCOMES:
McGill Pain Questionnaire-Dutch Language Version (MPQ-DLV)
Quebec Back Pain Disability Scale
Rand-36
EuroQoL (European Quality of Life Scale)
Costs (societal perspective)
Multidimensional Pain Inventory (MPI-DLV)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Terheggen, MD, Principal Investigator — Rijnstate Hospital; Maarten van Kleef, MD, PhD, Study Chair — UMC Maastricht
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands